CLINICAL TRIAL: NCT05877547
Title: A Phase 2b Randomized, Double-Blind, Placebo-Controlled, Multicenter Study to Evaluate the Efficacy and Safety of Efinopegdutide (MK-6024) in Adults With Precirrhotic Nonalcoholic Steatohepatitis
Brief Title: A Clinical Study of Efinopegdutide in Participants With Precirrhotic Nonalcoholic Steatohepatitis (NASH) (MK-6024-013)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 6024-013; 2022-502647-35-00 (Registry Identifier: EU CT); MK-6024-013 (Other: MSD); jRCT2031230187 (Registry Identifier: jRCT); U1111-1285-0933 (Registry Identifier: UTN)
Record Dates: First submitted 2023-05-17; First posted 2023-05-26 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Non-alcoholic Fatty Liver Disease; Fatty Liver, Nonalcoholic; NAFLD; Nonalcoholic Fatty Liver Disease; Nonalcoholic Steatohepatitis
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — semaglutide

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Efinopegdutide 4mg (Experimental): Efinopegdutide administered by subcutaneous (SC) injection once weekly for 52 weeks in a dose-escalation regimen of 2 mg for 4 weeks and 4mg for 48 weeks.
  Interventions: Drug: Efinopegdutide
- Efinopegdutide 7mg (Experimental): Efinopegdutide administered by SC injection once weekly for 52 weeks in a dose-escalation regimen of 2 mg for 4 weeks, 4 mg for 4 weeks, and 7 mg for 44 weeks.
  Interventions: Drug: Efinopegdutide
- Efinopegdutide 10mg (Experimental): Efinopegdutide administered by SC injection once weekly for 52 weeks in a dose-escalation regimen of 2 mg for 4 weeks, 4 mg for 4 weeks, 7 mg for 4 weeks, and 10 mg for 40 weeks.
  Interventions: Drug: Efinopegdutide
- Placebo (Placebo Comparator): Placebo administered by SC injection once weekly for 52 weeks
  Interventions: Drug: Placebo
- Semaglutide 2.4 mg (Active Comparator): Semaglutide administered by SC injection once weekly for 52 weeks in a dose-escalation regimen of 0.25 mg for 4 weeks, 0.5 mg for 4 weeks, 1.0 mg for 4 weeks, 1.7 mg for 4 weeks, and 2.4 mg for 36 weeks.
  Interventions: Drug: Semaglutide

INTERVENTIONS:
Drug: Efinopegdutide — Subcutaneous (SC) injection in dose-escalation regimens potentially including doses of 2 mg, 4 mg, 7 mg, and 10 mg
  Other Names: MK-6024; HM12525A; JNJ-64565111
  Arms: Efinopegdutide 10mg; Efinopegdutide 4mg; Efinopegdutide 7mg
Drug: Semaglutide — SC injection in a dose-escalation regimen of 0.25 mg, 0.5 mg, 1.0 mg, 1.7 mg, and 2.4 mg
  Other Names: Wegovy
  Arms: Semaglutide 2.4 mg
Drug: Placebo — SC injection of matching placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to learn how well efinopegdutide works compared to placebo in people who have non-alcoholic steatohepatitis (NASH). Researchers will also learn about the safety and benefit of efinopegdutide and how well people tolerate the medicine. The main goal of the study is to compare how many people taking efinopegdutide or placebo stop showing evidence of NASH without liver scarring getting worse.

ELIGIBILITY:
Inclusion Criteria:

* Histological confirmation of NASH, defined as NAFLD Activity Score (NAS) ≥4 with a score ≥1 point in each component (steatosis, ballooning, and lobular inflammation) AND NASH clinical research network (CRN) fibrosis score of Stage 2 or 3
* No history of Type 2 diabetes mellitus (T2DM) OR a history of T2DM with an A1C ≤9% that is controlled by diet or stable doses of antihyperglycemic agents (AHAs)
* Participants in South Korea are eligible between the ages of 19 to 80 years of age (inclusive)

Exclusion Criteria:

* History of liver disease other than NASH
* History or evidence of cirrhosis
* History of pancreatitis
* History of Type 1 diabetes mellitus (T1DM), diabetic ketoacidosis, or diabetes secondary to pancreatectomy
* History of a bariatric surgical procedure ≤5 years before study entry, or a known clinically significant gastric emptying abnormality
* Has significant systemic or major illnesses, including recent events (≤6 months before study entry) of congestive heart failure, unstable angina, myocardial infarction, arterial revascularization, stroke, or transient ischemic attack

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 381 (Actual)
Dates: Start 2023-06-23 (Actual); Primary Completion 2025-12-29 (Actual); Study Completion 2025-12-29 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants With Nonalcoholic Steatohepatitis (NASH) Resolution Without Worsening of Fibrosis At Week 52 | Week 52
  The NASH Clinical Research Network (CRN) scoring system evaluated by Blinded Independent Central Review (BICR) is used to assess treatment response. The NASH CRN scoring scales are: lobular inflammation score (0-3); hepatocyte ballooning score (0-2); steatosis score (0-3); and fibrosis score (0-4). NASH resolution is defined as a score of 0-1 for inflammation, 0 for ballooning, and any grade of steatosis.
Percentage of Participants Who Experienced an Adverse Event (AE) | Up to 60 weeks
  An adverse event (AE) is a health problem that happens or worsens during a study.
Percentage of Participants Discontinuing Study Medication Due to an AE | Up to 52 weeks
  An adverse event (AE) is a health problem that happens or worsens during a study.

SECONDARY OUTCOMES:
Percentage of Participants With ≥1 Stage Improvement in Fibrosis Without Worsening of Steatohepatitis At Week 52 | Week 52
  Participants will be assessed using the NASH CRN scoring system evaluated by BICR for ≥1-stage improvement in fibrosis without worsening of steatohepatitis. Fibrosis is scored from stage 0 to 4 where 0 = None, 1=Perisinusoidal OR periportal, 2=Perisinusoidal AND portal/periportal, 3= Bridging fibrosis, 4=Cirrhosis. No worsening of steatohepatitis is defined as no increase in the ballooning, inflammation, or steatosis scores.
Change from Baseline in Body Weight At Week 52 | Week 52
  Body weight (kg) will be measured using a standardized, digital scale. The percent change from baseline in body weight after 52 weeks will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (175):
- United States (42):
  - The Institute for Liver Health II dba Arizona Clinical Trial-The Institute for Liver Health ( Site 3, Chandler, Arizona
  - The Institute for Liver Health II dba Arizona Clinical Trials - Peoria ( Site 3289), Peoria, Arizona
  - The Institute for Liver Health II dba Arizona Liver Health-Tucson ( Site 3218), Tucson, Arizona
  - Del Sol Research Management, LLC ( Site 3211), Tucson, Arizona
  - Om Research - Apple Valley ( Site 3244), Apple Valley, California
  - Om Research LLC ( Site 3245), Camarillo, California
  - Velocity Clinical Research, Gardena ( Site 3225), Gardena, California
  - Velocity Clinical Research, Huntington Park ( Site 3217), Huntington Park, California
  - Velocity Clinical Research, San Diego ( Site 3226), La Mesa, California
  - Om Research LLC ( Site 3229), Lancaster, California
  - Velocity Clinical Research, Westlake ( Site 3216), Los Angeles, California
  - Velocity Clinical Research, Panorama City ( Site 3214), Panorama City, California
  - California Liver Research Institute ( Site 3232), Pasadena, California
  - Clinical Trials Research ( Site 3230), Sacramento, California
  - Excel Medical Clinical Trials ( Site 3246), Boca Raton, Florida
  - Synergy Healthcare ( Site 3286), Bradenton, Florida
  - Synergy Healthcare LLC ( Site 3290), Brandon, Florida
  - Top Medical Research ( Site 3209), Cutler Bay, Florida
  - Covenant Metabolic Specialists, LLC ( Site 3231), Fort Myers, Florida
  - Velocity Clinical Research, Hallandale Beach ( Site 3241), Hallandale, Florida
  - Indago Research & Health Center, Inc ( Site 3207), Hialeah, Florida
  - Sweet Hope Research Specialty, Inc-Research ( Site 3200), Hialeah, Florida
  - Florida Research Institute ( Site 3243), Lakewood Rch, Florida
  - Genoma Research Group ( Site 3242), Miami, Florida
  - Floridian Clinical Research, LLC ( Site 3203), Miami Lakes, Florida
  - Southeast Clinical Research Center ( Site 3288), Dalton, Georgia
  - Eagle Clinical Research ( Site 3233), Chicago, Illinois
  - University of Iowa ( Site 3213), Iowa City, Iowa
  - Kansas City Research Institute ( Site 3249), Kansas City, Missouri
  - The Machuca Foundation ( Site 3234), Las Vegas, Nevada
  - Velocity Clinical Research, Syracuse ( Site 3227), East Syracuse, New York
  - New York Gastroenterology Associates ( Site 3252), New York, New York
  - Velocity Clinical Research, Cincinnati ( Site 3237), Cincinnati, Ohio
  - Velocity Clinical Research, Providence ( Site 3222), East Greenwich, Rhode Island
  - Velocity Clinical Research, Austin ( Site 3235), Austin, Texas
  - South Texas Research Institute - Brownsville ( Site 3285), Brownsville, Texas
  - Velocity Clinical Research, Dallas ( Site 3220), Dallas, Texas
  - Houston Research Institute ( Site 3262), Houston, Texas
  - American Research Corporation ( Site 3202), San Antonio, Texas
  - Pinnacle Clinical Research ( Site 3284), San Antonio, Texas
  - Velocity Clinical Research, Salt Lake City ( Site 3223), West Jordan, Utah
  - Gastroenterology Consultants of Southwest Virginia ( Site 3282), Roanoke, Virginia
- Medizinische Universität Graz-Department of Internal Medicine ( Site 0302), Graz, Styria, Austria
- Belgium (3):
  - Antwerp University Hospital-Gastr-enterologie/hepatologie ( Site 3300), Edegem, Antwerpen
  - AZ Maria Middelares-Digestief Centrum ( Site 3301), Ghent, Oost-Vlaanderen
  - UZ Leuven-Hepatology ( Site 3302), Leuven, Vlaams-Brabant
- Canada (5):
  - Heritage Medical Research Clinic ( Site 0403), Calgary, Alberta
  - Vancouver General Hospital-Gastroenterology ( Site 0408), Vancouver, British Columbia
  - Toronto General Hospital ( Site 0402), Toronto, Ontario
  - McGill University Health Centre ( Site 0400), Montreal, Quebec
  - Diex Recherche Quebec Inc. ( Site 0409), Québec, Quebec
- Chile (3):
  - Enroll SpA ( Site 0501), Providencia, Region M. de Santiago
  - CECIM ( Site 0500), Santiago, Region M. de Santiago
  - Pontificia Universidad Catolica de Chile-CICUC ( Site 0502), Santiago, Region M. de Santiago
- China (9):
  - Beijing Youan Hospital ( Site 0602), Beijing, Beijing Municipality
  - Beijing Tsinghua Changgung Hospital ( Site 0606), Beijing, Beijing Municipality
  - Chongqing University Three Gorges Hospital ( Site 0607), Wanzhou, Chongqing Municipality
  - The First Affiliated Hospital, Sun Yat-sen University ( Site 0603), Guangzhou, Guangdong
  - Southern Medical University Nanfang Hospital ( Site 0601), Guangzhou, Guangdong
  - No. 2 Hospital of Nanjing ( Site 0605), Nanjing, Jiangsu
  - West China Hospital, Sichuan University ( Site 0611), Chengdu, Sichuan
  - Tianjin Second People's Hospital ( Site 0604), Tianjin, Tianjin Municipality
  - The First Affiliated Hospital of Wenzhou Medical University ( Site 0609), Wenzhou, Zhejiang
- Colombia (6):
  - Fundación Centro de Investigación Clínica CIC ( Site 0704), Medellín, Antioquia
  - Sociedad De Oncología y Hematología Del Cesar SAS ( Site 0708), Valledupar, Cesar Department
  - Fundacion Santa Fe de Bogota ( Site 0701), Bogotá, Cundinamarca
  - Solano & Terront Servicios Medicos - UNIENDO ( Site 0705), Bogotá, Cundinamarca
  - Oncomédica S.A.S ( Site 0702), Montería, Departamento de Córdoba
  - Fundación Valle del Lili ( Site 0700), Cali, Valle del Cauca Department
- Czechia (3):
  - KlinMed ( Site 0801), Prague, Praha 2
  - Krajská nemocnice Liberec ( Site 0800), Liberec
  - Vseobecna fakultni nemocnice v Praze ( Site 0802), Prague
- France (10):
  - Centre Hospitalier Universitaire de Nice - Hôpital l'Archet-Pôle de Référence Hépato Gastro-entérol, Nice, Alpes-Maritimes
  - CHU Bordeaux Haut-Leveque-Service d'Hépato-gastroentérologie ( Site 0904), Pessac, Aquitaine
  - Hôpital de la Croix Rousse-Centre de Recherche Clinique ( Site 0911), Lyon, Auvergne-Rhône-Alpes
  - centre hospitalier lyon sud-Endocrinologie, Diabète et Nutrition ( Site 0906), Pierre-Bénite, Auvergne-Rhône-Alpes
  - CHU Charles Nicolle ( Site 0910), Rouen, Haute-Normandie
  - Hôpital Beaujon-Hépatologie ( Site 0908), Clichy, Hauts-de-Seine
  - Centre Hospitalier Universitaire d'Angers-Hepato Gastroenterology ( Site 0900), Angers, Maine-et-Loire
  - Centre Hospitalier Universitaire Estaing ( Site 0913), Clermont-Ferrand, Puy-de-Dome
  - Hôpital Saint Antoine ( Site 0914), Paris
  - Hopitaux Universitaires Paris Centre-Hopital Cochin-Service HEPATOLOGIE- Recherche Clinique ( Site 0, Paris
- Prince of Wales Hospital ( Site 1000), Shatin, Hong Kong
- Hungary (2):
  - SYNEXUS Magyarország Kft. Eü. ( Site 1110), Budapest
  - Dél-Pesti Centrumkórház-Hepatologiai Szakrendekő ( Site 1102), Budapest
- Israel (7):
  - Barzilai Medical Center ( Site 1306), Ashkelon
  - Rambam Health Care Campus ( Site 1304), Haifa
  - Carmel Hospital ( Site 1305), Haifa
  - Shaare Zedek Medical Center-Liver Unit ( Site 1302), Jerusalem
  - Rabin Medical Center ( Site 1301), Petah Tikva
  - Sheba Medical Center ( Site 1300), Ramat Gan
  - Maccabi Health Services - Ramat Hasharon ( Site 1303), Ramat HaSharon
- Italy (5):
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS -Dipartimento di Medicina Interna e Gas, Rome, Lazio
  - Fondazione IRCCS Cà Granda Ospedale Maggiore Policlinico ( Site 1403), Milan, Lombardy
  - Humanitas-Medicina interna ed Epatologia ( Site 1400), Rozzano, Lombardy
  - A.O.U. Policlinico Paolo Giaccone-Dep. Of Internal Medicine and Specialistic ( Site 1402), Palermo, Sicily
  - Azienda Ospedaliero-Universitaria Città della Salute e della-S.C. Gastroenterologia U. ( Site 1401), Torino
- Japan (21):
  - Ehime University Hospital ( Site 1509), Tōon, Ehime
  - Kurume University Hospital ( Site 1504), Kurume, Fukuoka
  - Ogaki Municipal Hospital ( Site 1511), Ōgaki, Gifu
  - Sapporo Kosei General Hospital ( Site 1521), Sapporo, Hokkaido
  - Kagawa University Hospital ( Site 1515), Kita, Kagawa-ken
  - Kagawa Prefectural Central Hospital ( Site 1514), Takamatsu, Kagawa-ken
  - Toranomon Hospital Kajigaya ( Site 1502), Kawasaki, Kanagawa
  - Shinyurigaoka General Hospital ( Site 1518), Kawasaki, Kanagawa
  - St. Marianna University Hospital ( Site 1516), Kawasaki, Kanagawa
  - Yokohama City University Hospital ( Site 1505), Yokohama, Kanagawa
  - Shinshu University Hospital ( Site 1512), Matsumoto, Nagano
  - Nara Medical University Hospital ( Site 1513), Kashihara, Nara
  - Osaka Saiseikai Suita Hospital ( Site 1503), Suita, Osaka
  - Toranomon Hospital ( Site 1501), Minato-ku, Tokyo
  - Fukuiken Saiseikai Hospital ( Site 1507), Fukui
  - Gifu Municipal Hospital ( Site 1506), Gifu
  - University Hospital,Kyoto Prefectural University of Medicine ( Site 1519), Kyoto
  - Kawasaki Medical School General Medical Center ( Site 1508), Okayama
  - Osaka Metropolitan University Hospital ( Site 1520), Osaka
  - Saga University Hospital ( Site 1510), Saga
  - Japanese Red Cross Musashino Hospital ( Site 1517), Tokyo
- Mexico (8):
  - Medica Sur-Clinica de Enfermedades Digestivas y Obesidad ( Site 1603), Mexico City, Mexico City
  - Hospital Universitario "Dr. Jose Eleuterio Gonzalez" ( Site 1604), Monterrey, Nuevo León
  - Servicios de Oncología Médica Integral - Monterrey ( Site 1611), Monterrey, Nuevo León
  - ICARO Investigaciones en Medicina ( Site 1608), Chihuahua City
  - Centro de Investigación y Gastroenterología ( Site 1601), Cuauhtémoc
  - Centro de Investigación y Gastroenterología - S.C. ( Site 1609), Mexico City
  - Oaxaca Site Management Organization ( Site 1613), Oaxaca City
  - Centro de Investigacion Clinica de Oaxaca ( Site 1607), Oaxaca City
- Peru (3):
  - Centro de investigacion Clínica Trujillo ( Site 1802), Trujillo, La Libertad
  - CLINICA DELGADO-Clinical Research ( Site 1800), Miraflores, Lima region
  - Instituto Médico Soy Diabetico ( Site 1804), Piura
- Portugal (4):
  - Unidade Local de Saúde do Alto Ave - Hospital Senhora da Oliveira ( Site 1905), Guimarães, Braga District
  - Unidade Local de Saude Lisboa Ocidental - Hospital Egas Moniz ( Site 1906), Lisbon, Lisbon District
  - Unidade Local de Saude de Santa Maria - Hospital de Santa Maria ( Site 1904), Lisbon, Lisbon District
  - ULSAM - Hospital de Santa Luzia ( Site 1907), Viana do Castelo
- Puerto Rico (4):
  - ISIS CLINICAL RESEARCH CENTER ( Site 2006), Guaynabo
  - Pan American Center for Oncology Trials ( Site 2000), Rio Piedras
  - Klinical Investigations Group-Clinical Research ( Site 2001), San Juan
  - Latin Clinical Trial Center ( Site 2004), San Juan
- Singapore General Hospital ( Site 2188), Singapore, Central Singapore, Singapore
- South Korea (4):
  - Boramae Medical Center-Internal Medicine ( Site 2403), Dongjak-gu, Seoul
  - Inha University Hospital-Gastroenterolgy/Hepatology ( Site 2402), Incheon
  - Severance Hospital, Yonsei University Health System ( Site 2401), Seoul
  - Samsung Medical Center-Gastroenterology/Internal Medicine ( Site 2400), Seoul
- Spain (10):
  - Hospital Universitario Virgen de la Victoria-UGC Endocrinologia y nutricion ( Site 2506), Málaga, Andalusia
  - Hospital Universitario Marqués de Valdecilla-Gastroenterology and Hepatology ( Site 2505), Santander, Cantabria
  - Hospital General de Tomelloso-Aparato Digestivo ( Site 2514), Tomelloso, Ciudad Real
  - CHUAC-Complejo Hospitalario Universitario A Coruña-Endocrinología ( Site 2511), A Coruña, La Coruna
  - CHUS - Hospital Clinico Universitario ( Site 2503), Santiago de Compostela, La Coruna
  - Hospital Universitario Ramón y Cajal ( Site 2508), Madrid, Madrid, Comunidad de
  - Hospital Universitari Vall d'Hebron-Liver Unit - Department of Internal Medicine ( Site 2507), Barcelona
  - Hospital Universitario La Paz-HEPATOLOGIA ( Site 2509), Madrid
  - HOSPITAL UNIVERSITARIO PUERTA DE HIERRO MAJADAHONDA-Gastroenterologia y Hepatologia ( Site 2500), Madrid
  - HOSPITAL UNIVERSITARIO VIRGEN DEL ROCIO-Unidad de Ensayos Clínicos de Aparato Digestivo ( Site 2504), Seville
- Switzerland (3):
  - Cantonal Hospital St.Gallen-Klinik für Gastroenterologie / Hepatologie ( Site 2601), Sankt Gallen, Canton of St. Gallen
  - UniversitätsSpital Zürich-Gastroenterologie & Hepatologie ( Site 2603), Zurich, Canton of Zurich
  - Fondazione Epatocentro Ticino ( Site 2602), Lugano, Canton Ticino
- Taiwan (7):
  - Changhua Christian Hospital-Endocrinology and metabolism ( Site 2704), Changhua County, Changhua
  - Chiayi Christian Hospital ( Site 2707), Chiayi City, Chiayi
  - Taichung Veterans General Hospital ( Site 2703), Taichung
  - National Cheng Kung University Hospital-Liver Research team of National Cheng Kung University Hospi, Tainan
  - National Taiwan University Hospital-Internal Medicine ( Site 2700), Taipei
  - Taipei Veterans General Hospital-Division of Gastroenterology & Hepatology, Department of Medicine (, Taipei
  - Chang Gung Medical Foundation-Linkou Branch ( Site 2702), Taoyuan District
- Thailand (3):
  - Chulalongkorn University ( Site 2800), Bangkok, Bangkok
  - Faculty of Medicine Siriraj Hospital-Department of Medicine ( Site 2802), Bangkok, Bangkok
  - Maharaj Nakorn Chiang Mai Hospital ( Site 2801), Muang, Chiang Mai
- Turkey (Türkiye) (5):
  - Hacettepe Universite Hastaneleri-internal diseases ( Site 2901), Ankara
  - Bezmialem Vakf Üniversitesi-Gastroenterology ( Site 2903), Istanbul
  - T.C. Sağlik Bakanliği- Marmara Üniversitesi İstanbul Pendik -T.C. Sağlik Bakanliği- Marmara Ünivers, Istanbul
  - Dokuz Eylul Universitesi Hastanesi-Gastroenterology ( Site 2905), Izmir
  - Recep Tayyip Erdogan University Training and Research Hospital ( Site 2900), Rize
- United Kingdom (5):
  - Royal London Hospital ( Site 3003), London, England
  - King's College Hospital ( Site 3002), London, London, City of
  - Aberdeen Royal Infirmary-Department of Gastroenterology ( Site 3004), Aberdeen, Scotland
  - Queen Elizabeth Hospital Birmingham ( Site 3000), Birmingham, Warwickshire
  - St James's University Hospital ( Site 3005), Leeds

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26200&tenant=MT_MSD_9011